CLINICAL TRIAL: NCT00724789
Title: An Open-label, Observational Trial to Monitor the Incidence of Congenital Malformations in Infants of Women With an Ongoing Pregnancy After Controlled Ovarian Hyperstimulation Using Puregon® (recFSH)/Orgalutran® (Ganirelix) Followed by IVF/ICSI, or a Long Protocol With a GnRH Agonist as Historical Controls.
Brief Title: Monitor the Incidence of Congenital Malformations in Infants of Women Who Have Been Treated With Ganirelix (Orgalutran®)(Study 38644)(P05966)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05966; 38644
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy; Neonates
Keywords: Neonatal outcome; Congenital malformations; In-Vitro fertilization; Controlled ovarian stimulation; Follow-up
MeSH Terms: conditions — Congenital Abnormalities | interventions — ganirelix; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Observational Cohort: Subjects with an ongoing pregnancy after controlled ovarian stimulations with recombinant follicle stimulating hormone/ganirelix followed by in vitro fertilization or intra cytoplasmatic sperm injection.
  Interventions: Drug: ganirelix
- Historical Controls: Subjects with an ongoing pregnancy after controlled ovarian stimulations with recombinant follicle stimulating hormone in a long protocol with a gonadotropin releasing hormone agonist followed by IVF or ICSI
  Interventions: Drug: GnRH agonist

INTERVENTIONS:
Drug: ganirelix — Daily 0.25 mg ganirelix administered to prevent premature LH surges during COS in order to achieve a pregnancy
  Other Names: Orgalutran; Org 37462
  Groups: Observational Cohort
Drug: GnRH agonist — Long protocol of GnRH agonist administered to prevent premature LH surges during COS in order to achieve a pregnancy
  Groups: Historical Controls

SUMMARY:
The primary purpose of this study is to collect data on the incidence of congenital malformations in infants of women with an ongoing pregnancy after controlled ovarian stimulation with recombinant follicle stimulating hormone /ganirelix followed by in vitro fertilization (IVF) or intra cytoplasmatic sperm injection (ICSI), and to compare this incidence with that of a group of women who used a long protocol with a gonadotropin releasing hormone agonist as historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Puregon® (recFSH)/Orgalutran® group:

  * Women with a pregnancy of >= 16 weeks after Puregon® /Orgalutran® treatment for IVF or ICSI and ET of fresh embryos. Treatment is defined as having had at least one injection of Orgalutran®.
  * Women between 18 and 39 years of age (inclusive) at the day of hCG.
  * Women who are able and willing to sign informed consent.

Controls

* Infants (gestational age >=16 weeks) of women pregnant after COH using a GnRH agonist in a long protocol for IVF or ICSI and ET of fresh embryos.
* Infants of women between 18 and 39 years of age (inclusive) at the day of hCG.
* The most recent 1000 infants delivered prior to January 1, 2001.

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Single site study; A total of approximately 2000 infants born after IVF or ICSI: app. 1000 infants born after ongoing pregnancies resulting from COH including Puregon/Orgalutran treatment followed by IVF or ICSI and app. 1000 infants born after treatment with a long agonist protocol followed by IVF or ICSI as controls.
Sampling Method: Non-Probability Sample
Enrollment: 2066 (Actual)
Dates: Start 2000-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To collect data on the incidence of congenital malformations in infants of women with an ongoing pregnancy after controlled ovarian hyperstimulation. | In both cohorts a follow-up pediatric evaluation was scheduled within 6 months post-partum

REFERENCES:
- [Derived] Bonduelle M, Oberye J, Mannaerts B, Devroey P. Large prospective, pregnancy and infant follow-up trial assures the health of 1000 fetuses conceived after treatment with the GnRH antagonist ganirelix during controlled ovarian stimulation. Hum Reprod. 2010 Jun;25(6):1433-40. doi: 10.1093/humrep/deq072. Epub 2010 Apr 8. PMID 20378616